CLINICAL TRIAL: NCT05718648
Title: Pharmacokinetics, Safety and Tolerability of BI 1015550 Following Oral Administration in Male and Female Participants With Different Degrees of Renal Impairment (Severe and Moderate) as Compared With Individually Matched Male and Female Participants With Normal Renal Function (an Open-label, Non-randomised, Single Dose, Parallel, Individual-matched Design Trial)
Brief Title: A Study to Test How BI 1015550 is Taken up in the Blood of People With and Without Kidney Problems
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 1305-0025; 2022-003080-18 (EudraCT Number)
Record Dates: First submitted 2023-01-30; First posted 2023-02-08 (Actual); Results first posted 2025-11-28 (Actual); Last update posted 2025-11-28 (Actual); Status verified 2025-10

CONDITIONS: Renal Insufficiency; Healthy
MeSH Terms: conditions — Renal Insufficiency | interventions — BI 1015550

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- BI 1015550 Severe renal impairment (Experimental): Participants with severe renal impairment (estimated glomerular filtration rate (eGFR)) according to Chronic Kidney Disease Epidemiology Collaboration 15-29 milliliter(mL)/minute(min)/1.73 meter(m)²), and not requiring dialysis, administered orally one film-coated tablet of 18 milligram (mg) of BI 1015550 with 240 mL of water after an overnight fast of at least 10 hours (h).
  Interventions: Drug: BI 1015550
- BI 1015550 Moderate renal impairment (Experimental): Participants with moderate renal impairment (eGFR 30-59 mL/min/1.73 m²) administered orally one film-coated tablet of 18 mg of BI 1015550 with 240 mL of water after an overnight fast of at least 10 h.
  Interventions: Drug: BI 1015550
- BI 1015550 Normal renal function (Experimental): Participants with normal renal function (eGFR ≥90 mL/min/1.73 m²) administered orally one film-coated tablet of 18 mg of BI 1015550 with 240 mL of water after an overnight fast of at least 10 h.
  Participants with normal renal function were individually matched by age (± 10 years), gender, weight (± 15%), and race to the participants with renal impairment. Each participant with normal renal function could be matched to one participant with moderate renal impairment and to one participant with severe renal impairment.
  Interventions: Drug: BI 1015550

INTERVENTIONS:
Drug: BI 1015550 — BI 1015550
  Other Names: Nerandomilast; JASCAYD®

SUMMARY:
This study is open to adults aged 18 years and older. People without kidney problems and people who have moderate or severe kidney problems can join the study.

The purpose of this study is to find out how a medicine called BI 1015550 is taken up in the blood of people with and without kidney problems. Kidney problems may change how a medicine is taken up in the blood. All participants take a single tablet of BI 1015550.

Participants are in the study for about 2 weeks. During this time, they visit the study site 6 times. On the second visit, participants stay overnight at the study site for 4 nights. At the visits, doctors take blood samples to measure the levels of BI 1015550 in participants' blood. Then they compare the results between the groups of participants with and without kidney problems. The doctors also check participants' health and take note of any unwanted effects.

ELIGIBILITY:
Inclusion Criteria:

Inclusion criteria applying to all participants:

* Male or female participants
* Age of 18-79 years (inclusive)
* Body mass index (BMI) of 18.5 to 35.0 kg/m2 (inclusive)
* Signed and dated written informed consent in accordance with International Council for Harmonisation-Good Clinical Practice (ICH-GCP) and local legislation prior to admission to the trial
* Male participants are not required to use contraception
* Women of child-bearing potential (WOCBP) are allowed to participate provided they use a highly effective contraception from at least 30 days before the administration of trial medication until 7 days after trial completion.

Of note, oral hormonal contraceptives are not considered as highly effective in this study due to the potential CYP3A induction by BI 1015550. Therefore, the following methods of contraception are considered adequate for female participants of childbearing potential:

* Use of combined (oestrogen and progestogen containing) hormonal contraception that prevents ovulation (oral, intravaginal or transdermal), plus condom
* Use of progestogen-only hormonal contraception that inhibits ovulation (only injectables or implants), plus condom
* Use of intrauterine device (IUD) or intrauterine hormone-releasing system (IUS)
* Sexually abstinent
* A vasectomised sexual partner who received medical assessment of the surgical success (documented absence of sperm) and provided that partner is the sole sexual partner of the trial participant.

Female participants are not considered to be of childbearing potential if they are either surgically sterilised (including hysterectomy) or postmenopausal, defined as no menses for 1 year without an alternative medical cause (in questionable cases, a blood sample with levels of Follicle stimulating hormone (FSH) above 40 units per liter (U/L) and oestradiol below 30 nanograms/liter (ng/L) is confirmatory).

Further inclusion criteria apply.

Exclusion Criteria:

Exclusion criteria applying to all participants:

* Any evidence of a concomitant disease assessed as clinically relevant by the investigator
* Cholecystectomy or other surgery of the gastrointestinal (GI) tract that could interfere with the pharmacokinetics of the trial medication (except appendectomy or simple hernia repair)
* Diseases of the central nervous system (CNS) (including but not limited to any kind of seizures or stroke), and other relevant neurological or psychiatric disorders (including but not limited to major depressive disorder)
* History of relevant orthostatic hypotension, fainting spells, or blackouts
* Relevant chronic or acute infections
* Any documented active or suspected malignancy or history of malignancy within 5 years prior to screening, except appropriately treated basal cell carcinoma of the skin or squamous cell carcinoma in situ of the skin or in situ carcinoma of uterine cervix
* History of relevant allergy or hypersensitivity (including allergy to the trial medication or its excipients)
* Use of drugs within 30 days (or 5 of their half-lives, whichever is longer) of planned administration of trial medication that might reasonably influence the results of the trial (including drugs that cause QT/QT interval corrected for heart rate (QTc) interval prolongation) Further exclusion criteria apply.

Ages: 18 Years to 79 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 26 (Actual)
Dates: Start 2023-02-09 (Actual); Primary Completion 2023-08-15 (Actual); Study Completion 2023-08-15 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- CRS Clinical Research Services Kiel GmbH, Kiel, Germany

IPD SHARING:
Plan to Share IPD: No
Clinical studies sponsored by Boehringer Ingelheim, phases I to IV, interventional and non-interventional, are in scope for sharing of the raw clinical study data and clinical study documents. Exceptions might apply, e.g. studies in products where Boehringer Ingelheim is not the license holder; studies regarding pharmaceutical formulations and associated analytical methods, and studies pertinent to pharmacokinetics using human biomaterials; studies conducted in a single center or targeting rare diseases (in case of low number of patients and therefore limitations with anonymization).
  For more details refer to:
  https://www.mystudywindow.com/msw/datatransparency

REFERENCES:
- See also: Related Info — https://www.mystudywindow.com

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This Phase I trial applied a non-randomised, parallel matched-group design and included participants with moderate or severe renal impairment and participants with normal renal function (matched controls to participants with renal impairment). All trial participants received one 18 milligram BI 1015550 tablet, administered in the fasting state.
Pre-assignment Details: All participants were screened for eligibility prior to participation in the trial. Participants attended a specialist site which ensured that the participants strictly met all inclusion and none of the exclusion criteria. Participants were not to be entered in the trial if any of the entry criteria were violated.
Period: Overall Study
Arm/Group | BI 1015550 Severe renal impairment | BI 1015550 Moderate renal impairment | BI 1015550 Normal renal function
Started | 8 | 8 | 10
Treated | 8 | 8 | 10
Completed | 8 | 8 | 10
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Treated set (TS): included all participants who received trial medication.
Groups:
- Total: Total of all reporting groups
Arm/Group | BI 1015550 Severe Renal Impairment | BI 1015550 Moderate Renal Impairment | BI 1015550 Normal Renal Function | Total
Number analyzed (Participants) | 8 | 8 | 10 | 26
Age, Continuous [Mean (Standard Deviation); unit: Years] | 66.4 (12.3) | 65.3 (10.3) | 60.7 (11.9) | 63.8 (11.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 | 3 | 4 | 11
  Male | 4 | 5 | 6 | 15
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 0
  White | 8 | 8 | 10 | 26
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Area Under the Concentration-time Curve of R-BI 1015550 in Plasma Over the Time Interval From 0 to the Last Quantifiable Data Point (AUC0-tz)
Description: Area under the concentration-time curve of R-BI 1015550 (the pharmacologically active R-enantiomer, measured by a chiral assay) in plasma over the time interval from 0 to the last quantifiable data point (AUC0-tz) is reported.
  Geometric least square mean (adjusted geometric mean) and adjusted geometric standard error were calculated using an analysis of variance (ANOVA) model on the logarithmic scale. The pharmacokinetic (PK) endpoints were log-transformed (natural logarithm) prior to fitting the ANOVA model. This model included effects accounting for the following sources of variation: 'degree of renal impairment' as fixed effect as well as 'matched pair' as random effect. These quantities were then back-transformed to the original scale.
  The ratio of adjusted geometric means is calculated with patients with renal impairment as test groups and their respective matched controls as reference groups.
Time Frame: Within 2 hours (h) prior to drug administration and 0.5, 0.75, 1, 1.25, 1.5, 1.75, 2, 2.5, 3, 4, 6, 8, 10, 12, 14, 24, 36, 48, 72, 96, 120 and 144 h after drug administration.
Population: Pharmacokinetic parameter analysis set (PKS): included all participants in the treated set (TS) who provided at least one PK endpoint that was defined as primary or secondary and that was not excluded due to a protocol deviation relevant to the evaluation of PK or due to PK non-evaluability. A participant was to be included in the PKS, even if he/she contributed only 1 PK parameter value to the statistical assessment.
Measure: Geometric Least Squares Mean (Standard Error); unit: hour*nanomole/Liter
Groups:
- BI 1015550 Normal renal function matched to severe renal impairment: Participants with normal renal function (eGFR ≥90 mL/min/1.73 m²) administered orally one film-coated tablet of 18 mg of BI 1015550 with 240 mL of water after an overnight fast of at least 10 h.
  Participants with normal renal function were individually matched by age (± 10 years), gender, weight (± 15%), and race to participants with severe renal impairment.
- BI 1015550 Normal renal function matched to moderate renal impairment: Participants with normal renal function (eGFR ≥90 mL/min/1.73 m²) administered orally one film-coated tablet of 18 mg of BI 1015550 with 240 mL of water after an overnight fast of at least 10 h.
  Participants with normal renal function were individually matched by age (± 10 years), gender, weight (± 15%), and race to participants with moderate renal impairment.
Arm/Group | BI 1015550 Severe renal impairment | BI 1015550 Normal renal function matched to severe renal impairment | BI 1015550 Moderate renal impairment | BI 1015550 Normal renal function matched to moderate renal impairment
Number analyzed (Participants) | 8 | 8 | 8 | 8
hour*nanomole/Liter | 3347.73 (NA) — Adjusted geometric standard error = 1.18 | 2590.32 (NA) — Adjusted geometric standard error = 1.18 | 3141.86 (NA) — Adjusted geometric standard error = 1.19 | 2285.92 (NA) — Adjusted geometric standard error = 1.19
Statistical Analysis 1: Comparison: BI 1015550 Severe renal impairment vs BI 1015550 Normal renal function matched to severe renal impairment; Ratio of adjusted geometric means was calculated using an analysis of variance (ANOVA) model on the logarithmic scale. The pharmacokinetic (PK) endpoints were log-transformed (natural logarithm) prior to fitting the ANOVA model. This model included effects accounting for the following sources of variation: 'degree of renal impairment' as fixed effect as well as 'matched pair' as random effect. These quantities were then back-transformed to the original scale; Test type: Other; Ratio of adjusted geometric means [%] = 129.24, 90% CI 2-sided [91.62 to 182.31] — Ratio [%] = (adjusted geometric mean of severe renal impairment / adjusted geometric mean matching control)*100. Intra-matched pair geometric coefficient of variation (gCV) [%] = 37.5
Statistical Analysis 2: Comparison: BI 1015550 Moderate renal impairment vs BI 1015550 Normal renal function matched to moderate renal impairment; [analysis description as in outcome 1, analysis 1]; Test type: Other; Ratio of adjusted geometric means [%] = 137.44, 90% CI 2-sided [89.06 to 212.12] — Ratio [%] = (adjusted geometric mean of moderate renal impairment / adjusted geometric mean matching control)*100. Intra-matched pair geometric coefficient of variation (gCV) [%] = 52.4

2. Primary Outcome: Area Under the Concentration-time Curve of BI 1015550 in Plasma Over the Time Interval From 0 to the Last Quantifiable Data Point (AUC0-tz)
Description: Area under the concentration-time curve of BI 1015550 (mixture of R-(pharmacologically active) and S-(pharmacologically inactive) enantiomers, measured by a non-chiral assay) in plasma over the time interval from 0 to the last quantifiable data point (AUC0-tz) is reported.
  Geometric least square mean (adjusted geometric mean) and adjusted geometric standard error were calculated using an analysis of variance (ANOVA) model on the logarithmic scale. The pharmacokinetic (PK) endpoints were log-transformed (natural logarithm) prior to fitting the ANOVA model. This model included effects accounting for the following sources of variation: 'degree of renal impairment' as fixed effect as well as 'matched pair' as random effect. These quantities were then back-transformed to the original scale.
  The ratio of adjusted geometric means is calculated with patients with renal impairment as test groups and their respective matched controls as reference groups.
Time Frame: as for outcome 1
Population: Pharmacokinetic parameter analysis set (PKS): included all participants in the TS who provided at least one PK endpoint that was defined as primary or secondary and that was not excluded due to a protocol deviation relevant to the evaluation of PK or due to PK non-evaluability. A participant was to be included in the PKS, even if he/she contributed only 1 PK parameter value to the statistical assessment.
Measure: Geometric Least Squares Mean (Standard Error); unit: hour*nanomole/Liter
Arm/Group | BI 1015550 Severe renal impairment | BI 1015550 Normal renal function matched to severe renal impairment | BI 1015550 Moderate renal impairment | BI 1015550 Normal renal function matched to moderate renal impairment
Number analyzed (Participants) | 8 | 8 | 8 | 8
hour*nanomole/Liter | 4367.05 (NA) — Adjusted geometric standard error = 1.17 | 3312.70 (NA) — Adjusted geometric standard error = 1.17 | 3841.47 (NA) — Adjusted geometric standard error = 1.16 | 3014.58 (NA) — Adjusted geometric standard error = 1.16
Statistical Analysis 1: Comparison: BI 1015550 Severe renal impairment vs BI 1015550 Normal renal function matched to severe renal impairment; [analysis description as in outcome 1, analysis 1]; Test type: Other; Ratio of adjusted geometric means [%] = 131.83, 90% CI 2-sided [93.32 to 186.22] — Ratio [%] = (adjusted geometric mean of severe renal impairment / adjusted geometric mean matching control)*100. Intra-matched pair geometric coefficient of variation (gCV) [%] = 37.7
Statistical Analysis 2: Comparison: BI 1015550 Moderate renal impairment vs BI 1015550 Normal renal function matched to moderate renal impairment; [analysis description as in outcome 1, analysis 1]; Test type: Other; Ratio of adjusted geometric means [%] = 127.43, 90% CI 2-sided [85.92 to 188.99] — Ratio [%] = (adjusted geometric mean of moderate renal impairment / adjusted geometric mean matching control)*100. Intra-matched pair geometric coefficient of variation (gCV) [%] = 43.5

3. Primary Outcome: Maximum Measured Concentration of R-BI 1015550 in Plasma (Cmax)
Description: Maximum measured concentration of R-BI 1015550 (the pharmacologically active R-enantiomer, measured by a chiral assay) in plasma (Cmax) is reported.
  Geometric least square mean (adjusted geometric mean) and adjusted geometric standard error were calculated using an analysis of variance (ANOVA) model on the logarithmic scale. The pharmacokinetic (PK) endpoints were log-transformed (natural logarithm) prior to fitting the ANOVA model. This model included effects accounting for the following sources of variation: 'degree of renal impairment' as fixed effect as well as 'matched pair' as random effect. These quantities were then back-transformed to the original scale.
  The ratio of adjusted geometric means is calculated with patients with renal impairment as test groups and their respective matched controls as reference groups.
Time Frame: as for outcome 1
Population: as for outcome 2
Measure: Geometric Least Squares Mean (Standard Error); unit: nanomole/Liter
Arm/Group | BI 1015550 Severe renal impairment | BI 1015550 Normal renal function matched to severe renal impairment | BI 1015550 Moderate renal impairment | BI 1015550 Normal renal function matched to moderate renal impairment
Number analyzed (Participants) | 8 | 8 | 8 | 8
nanomole/Liter | 399.46 (NA) — Adjusted geometric standard error = 1.12 | 464.19 (NA) — Adjusted geometric standard error = 1.12 | 367.36 (NA) — Adjusted geometric standard error = 1.24 | 380.43 (NA) — Adjusted geometric standard error = 1.24
Statistical Analysis 1: Comparison: BI 1015550 Severe renal impairment vs BI 1015550 Normal renal function matched to severe renal impairment; [analysis description as in outcome 1, analysis 1]; Test type: Other; Ratio of adjusted geometric means [%] = 86.06, 90% CI 2-sided [64.88 to 114.15] — Ratio [%] = (adjusted geometric mean of severe renal impairment / adjusted geometric mean matching control)*100. Intra-matched pair geometric coefficient of variation (gCV) [%] = 30.5
Statistical Analysis 2: Comparison: BI 1015550 Moderate renal impairment vs BI 1015550 Normal renal function matched to moderate renal impairment; [analysis description as in outcome 1, analysis 1]; Test type: Other; Ratio of adjusted geometric means [%] = 96.57, 90% CI 2-sided [56.80 to 164.16] — Ratio [%] = (adjusted geometric mean of moderate renal impairment / adjusted geometric mean matching control)*100. Intra-matched pair geometric coefficient of variation (gCV) [%] = 66.2

4. Primary Outcome: Maximum Measured Concentration of BI 1015550 in Plasma (Cmax)
Description: Maximum measured concentration of BI 1015550 (mixture of R-(pharmacologically active) and S-(pharmacologically inactive) enantiomers, measured by a non-chiral assay) in plasma (Cmax) is reported.
  Geometric least square mean (adjusted geometric mean) and adjusted geometric standard error were calculated using an analysis of variance (ANOVA) model on the logarithmic scale. The pharmacokinetic (PK) endpoints were log-transformed (natural logarithm) prior to fitting the ANOVA model. This model included effects accounting for the following sources of variation: 'degree of renal impairment' as fixed effect as well as 'matched pair' as random effect. These quantities were then back-transformed to the original scale.
  The ratio of adjusted geometric means is calculated with patients with renal impairment as test groups and their respective matched controls as reference groups.
Time Frame: as for outcome 1
Population: as for outcome 2
Measure: Geometric Least Squares Mean (Standard Error); unit: nanomole/Liter
Arm/Group | BI 1015550 Severe renal impairment | BI 1015550 Normal renal function matched to severe renal impairment | BI 1015550 Moderate renal impairment | BI 1015550 Normal renal function matched to moderate renal impairment
Number analyzed (Participants) | 8 | 8 | 8 | 8
nanomole/Liter | 404.41 (NA) — Adjusted geometric standard error = 1.13 | 486.36 (NA) — Adjusted geometric standard error = 1.13 | 359.75 (NA) — Adjusted geometric standard error = 1.25 | 397.56 (NA) — Adjusted geometric standard error = 1.25
Statistical Analysis 1: Comparison: BI 1015550 Severe renal impairment vs BI 1015550 Normal renal function matched to severe renal impairment; [analysis description as in outcome 1, analysis 1]; Test type: Other; Ratio of adjusted geometric means [%] = 83.15, 90% CI 2-sided [60.91 to 113.51] — Ratio [%] = (adjusted geometric mean of severe renal impairment / adjusted geometric mean matching control)*100. Intra-matched pair geometric coefficient of variation (gCV) [%] = 33.8
Statistical Analysis 2: Comparison: BI 1015550 Moderate renal impairment vs BI 1015550 Normal renal function matched to moderate renal impairment; [analysis description as in outcome 1, analysis 1]; Test type: Other; Ratio of adjusted geometric means [%] = 90.49, 90% CI 2-sided [52.40 to 156.26] — Ratio [%] = (adjusted geometric mean of moderate renal impairment / adjusted geometric mean matching control)*100. Intra-matched pair geometric coefficient of variation (gCV) [%] = 68.5

5. Secondary Outcome: Area Under the Concentration-time Curve of R-BI 1015550 in Plasma Over the Time Interval From 0 Extrapolated to Infinity (AUC0-∞)
Description: Area under the concentration-time curve of R-BI 1015550 (the pharmacologically active R-enantiomer, measured by a chiral assay) in plasma over the time interval from 0 extrapolated to infinity (AUC0-∞) is reported.
  Geometric least square mean (adjusted geometric mean) and adjusted geometric standard error were calculated using an analysis of variance (ANOVA) model on the logarithmic scale. The pharmacokinetic (PK) endpoints were log-transformed (natural logarithm) prior to fitting the ANOVA model. This model included effects accounting for the following sources of variation: 'degree of renal impairment' as fixed effect as well as 'matched pair' as random effect. These quantities were then back-transformed to the original scale.
  The ratio of adjusted geometric means is calculated with patients with renal impairment as test groups and their respective matched controls as reference groups.
Time Frame: as for outcome 1
Population: Pharmacokinetic parameter analysis set (PKS): included all participants in the TS who provided at least one PK endpoint that was defined as primary or secondary and that was not excluded due to a protocol deviation relevant to the evaluation of PK or due to PK non-evaluability. A participant was to be included in the PKS, even if he/she contributed only 1 PK parameter value to the statistical assessment. Only participants with available PK data are included in the analysis.
Measure: Geometric Least Squares Mean (Standard Error); unit: hour*nanomole/Liter
Arm/Group | BI 1015550 Severe renal impairment | BI 1015550 Normal renal function matched to severe renal impairment | BI 1015550 Moderate renal impairment | BI 1015550 Normal renal function matched to moderate renal impairment
Number analyzed (Participants) | 7 | 8 | 8 | 8
hour*nanomole/Liter | 3391.98 (NA) — Adjusted geometric standard error = 1.20 | 2638.63 (NA) — Adjusted geometric standard error = 1.18 | 3177.31 (NA) — Adjusted geometric standard error = 1.19 | 2333.59 (NA) — Adjusted geometric standard error = 1.19
Statistical Analysis 1: Comparison: BI 1015550 Severe renal impairment vs BI 1015550 Normal renal function matched to severe renal impairment; [analysis description as in outcome 1, analysis 1]; Test type: Other; Ratio of adjusted geometric means [%] = 128.55, 90% CI 2-sided [87.42 to 189.02] — Ratio [%] = (adjusted geometric mean of severe renal impairment / adjusted geometric mean matching control)*100. Intra-matched pair geometric coefficient of variation (gCV) [%] = 39.8
Statistical Analysis 2: Comparison: BI 1015550 Moderate renal impairment vs BI 1015550 Normal renal function matched to moderate renal impairment; [analysis description as in outcome 1, analysis 1]; Test type: Other; Ratio of adjusted geometric means [%] = 136.16, 90% CI 2-sided [88.41 to 209.69] — Ratio [%] = (adjusted geometric mean of moderate renal impairment / adjusted geometric mean matching control)*100. Intra-matched pair geometric coefficient of variation (gCV) [%] = 52.1

6. Secondary Outcome: Area Under the Concentration-time Curve of BI 1015550 in Plasma Over the Time Interval From 0 Extrapolated to Infinity (AUC0-∞)
Description: Area under the concentration-time curve of BI 1015550 (mixture of R-(pharmacologically active) and S-(pharmacologically inactive) enantiomers, measured by a non-chiral assay) in plasma over the time interval from 0 extrapolated to infinity (AUC0-∞) is reported.
  Geometric least square mean (adjusted geometric mean) and adjusted geometric standard error were calculated using an analysis of variance (ANOVA) model on the logarithmic scale. The pharmacokinetic (PK) endpoints were log-transformed (natural logarithm) prior to fitting the ANOVA model. This model included effects accounting for the following sources of variation: 'degree of renal impairment' as fixed effect as well as 'matched pair' as random effect. These quantities were then back-transformed to the original scale.
  The ratio of adjusted geometric means is calculated with patients with renal impairment as test groups and their respective matched controls as reference groups.
Time Frame: as for outcome 1
Population: as for outcome 5
Measure: Geometric Least Squares Mean (Standard Error); unit: hour*nanomole/Liter
Arm/Group | BI 1015550 Severe renal impairment | BI 1015550 Normal renal function matched to severe renal impairment | BI 1015550 Moderate renal impairment | BI 1015550 Normal renal function matched to moderate renal impairment
Number analyzed (Participants) | 7 | 8 | 8 | 8
hour*nanomole/Liter | 4280.84 (NA) — Adjusted geometric standard error = 1.19 | 3423.14 (NA) — Adjusted geometric standard error = 1.18 | 3941.06 (NA) — Adjusted geometric standard error = 1.16 | 3112.82 (NA) — Adjusted geometric standard error = 1.16
Statistical Analysis 1: Comparison: BI 1015550 Severe renal impairment vs BI 1015550 Normal renal function matched to severe renal impairment; [analysis description as in outcome 1, analysis 1]; Test type: Other; Ratio of adjusted geometric means [%] = 125.06, 90% CI 2-sided [85.27 to 183.40] — Ratio [%] = (adjusted geometric mean of severe renal impairment / adjusted geometric mean matching control)*100. Intra-matched pair geometric coefficient of variation (gCV) [%] = 39.6
Statistical Analysis 2: Comparison: BI 1015550 Moderate renal impairment vs BI 1015550 Normal renal function matched to moderate renal impairment; [analysis description as in outcome 1, analysis 1]; Test type: Other; Ratio of adjusted geometric means [%] = 126.61, 90% CI 2-sided [85.30 to 187.92] — Ratio [%] = (adjusted geometric mean of moderate renal impairment / adjusted geometric mean matching control)*100. Intra-matched pair geometric coefficient of variation (gCV) [%] = 43.6

ADVERSE EVENTS:
Time Frame: From the time of drug administration, until the end of the on-treatment period, up to 7 days. All-cause mortality was recorded from the time of drug administration until the end of trial, up to 2 weeks.
Description: Treated set included all participants who received trial medication. Adverse events are reported by impairment group according to the Statistical Analysis Plan. The sum of matched controls to the renal impairment groups (16) does not match the number of total participants with normal renal function (10), because 6 controls were matched to 1 participant with moderate renal impairment and to 1 participant with severe renal impairment.
Groups:
- BI 1015550 Severe renal impairment: Participants with severe renal impairment (eGFR according to Chronic Kidney Disease Epidemiology Collaboration 15-29 mL/min/1.73 m²), and not requiring dialysis, administered orally one film-coated tablet of 18 mg of BI 1015550 with 240 mL of water after an overnight fast of at least 10 h.
- BI 1015550 Normal renal function matched to moderate renal impairment: Participants with normal renal function (estimated glomerular filtration rate (eGFR) ≥90 milliliter(mL)/minute(min)/1.73 meter(m)²) administered orally one film-coated tablet of 18 mg of BI 1015550 with 240 mL of water after an overnight fast of at least 10 h.
  Participants with normal renal function were individually matched by age (± 10 years), gender, weight (± 15%), and race to participants with moderate renal impairment.
Arm/Group | BI 1015550 Severe renal impairment | BI 1015550 Normal renal function matched to severe renal impairment | BI 1015550 Moderate renal impairment | BI 1015550 Normal renal function matched to moderate renal impairment
All-Cause Mortality (participants affected / at risk) | 0/8 | 0/8 | 0/8 | 0/8
Serious Adverse Events (participants affected / at risk) | 0/8 | 0/8 | 0/8 | 0/8
Other Adverse Events (participants affected / at risk) | 4/8 | 3/8 | 2/8 | 3/8
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | BI 1015550 Severe renal impairment (N=8) | BI 1015550 Normal renal function matched to severe renal impairment (N=8) | BI 1015550 Moderate renal impairment (N=8) | BI 1015550 Normal renal function matched to moderate renal impairment (N=8)
Hypertension (Vascular disorders) | 2 | 0 | 0 | 0
Haematoma (Vascular disorders) | 0 | 1 | 0 | 1
Diarrhoea (Gastrointestinal disorders) | 0 | 0 | 1 | 0
COVID-19 (Infections and infestations) | 1 | 0 | 0 | 0
Nasopharyngitis (Infections and infestations) | 1 | 0 | 0 | 0
Contusion (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0
Lipase increased (Investigations) | 0 | 1 | 1 | 1
Dizziness (Nervous system disorders) | 1 | 0 | 0 | 0
Headache (Nervous system disorders) | 1 | 1 | 1 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Boehringer Ingelheim (BI) acknowledges that investigators have the right to publish the study results. Investigators shall provide BI with a copy of any publication or presentation for review prior to any submission. Such review will be done with regard to proprietary information, information related to patentable inventions, medical, scientific, and statistical accuracy within 60 days. BI may request a delay of the publication in order to protect BI's intellectual property rights.

DOCUMENTS (2):
  • Study Protocol (2023-01-10): https://cdn.clinicaltrials.gov/large-docs/48/NCT05718648/Prot_000.pdf
  • Statistical Analysis Plan (2023-09-18): https://cdn.clinicaltrials.gov/large-docs/48/NCT05718648/SAP_001.pdf